CLINICAL TRIAL: NCT04717258
Title: Do Safe and Well Visits Delivered by the Fire and Rescue Service Reduce Falls and Improve Quality of Life Among Older People? A Randomised Controlled Trial
Brief Title: Safe and Well Visits by the Fire and Rescue Service to Prevent Falls and Improve Quality of Life in Older People
Acronym: FIREFLI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Caroline Fairhurst (Other)
Collaborators: Humberside Fire and Rescue Service (Unknown); Leicestershire Partnership NHS Trust (Other); University of Nottingham (Other); Kent Fire and Rescue Service (Unknown); James Cook University, Queensland, Australia (Other); Queensland Health (Other Government)
Responsible Party: Sponsor-Investigator, Caroline Fairhurst, Senior statistician, University of York
Organization: University of York (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIREFLI Trial Protocol v6.0
Record Dates: First submitted 2020-12-09; First posted 2021-01-22 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Accidental Fall; Quality of Life; Aged
MeSH Terms: interventions — Fires

STUDY DESIGN:
Intervention Model Description: This study consists of a two-arm main trial, with two embedded two-arm SWATs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Main FIREFLI trial: Intervention arm (Experimental): Usual care from healthcare professionals; falls prevention leaflet; Safe and Well Visits (SWVs) offered by the Fire and Rescue Service (FRS) (either a firefighter, day duty safety advocate or home safety officer) once randomised.
  Interventions: Other: Fire and Rescue Service Safe and Well Visit
- Main FIREFLI trial: Control arm (No Intervention): Usual care from healthcare professionals; falls prevention leaflet; Safe and Well Visits (SWVs) by the Fire and Rescue Service (FRS) (either a firefighter, day duty safety advocate or home safety officer offered 12 months post-randomisation)
- Recruitment SWAT: Self-Determination Theory informed invitation letter (Experimental): The recruitment pack to take part in the FIREFLI study will include an invitation letter informed by Self-Determination Theory.
  Interventions: Other: Self-Determination Theory informed trial invitation letter
- Recruitment SWAT: Standard invitation letter (No Intervention): The recruitment pack to take part in the FIREFLI study will include the University of York, York Trials Unit's standard invitation letter
- Retention SWAT: Pen arm (Experimental): A pen (which has the University of York logo on it) will be included with the first four-month reminder questionnaire.
  Interventions: Other: Pen included with reminder questionaire
- Retention SWAT: No pen (No Intervention): No pen will be included with the four-month reminder questionnaire.

INTERVENTIONS:
Other: Fire and Rescue Service Safe and Well Visit — Safe and Well Visits by the Fire and Rescue Service to prevent falls and improve quality of life in an older population
  Arms: Main FIREFLI trial: Intervention arm
Other: Self-Determination Theory informed trial invitation letter — Invitation letter to take part in the FIREFLI study informed by Self-Determination Theory
  Arms: Recruitment SWAT: Self-Determination Theory informed invitation letter
Other: Pen included with reminder questionaire — A pen will be included with the four-month reminder questionnaire.
  Arms: Retention SWAT: Pen arm

SUMMARY:
FIREFLI is a large, pragmatic, individually randomised, controlled trial with embedded economic and qualitative evaluations. The aim of the research is to see whether Safe and Well Visits delivered by the Fire and Rescue Service will lead to a reduction in the number of falls and an improvement in health-related quality of life in older people. It will also look at the cost-effectiveness of the intervention and explore the acceptability of the Safe and Well Visits to older people and the Fire and Rescue Service.

The investigators will recruit 1156 participants, randomly divided into two equal groups. One group (the intervention group) will receive the Safe and Well Visit at the beginning of the study and the other group (the control group) will receive the visit at the end of the study.

The investigators will collect the number of falls people have using monthly falls calendars and follow up other outcomes by questionnaires at four, eight and 12 months post-randomisation. The investigators will also undertake interviews with some participants and with Fire and Rescue Service staff to explore experiences around the Safe and Well Visits.

Two Studies within a Trial (SWAT) will be carried out to investigate more efficient ways of running trials. The first will test if using a recruitment invitation letter informed by Self-Determination Theory will increase the number of participants who take part in the study. The second will test if including a pen with the reminder four-month questionnaire will increase the number of postal questionnaires returned to the study team.

DETAILED DESCRIPTION:
The Fire and Rescue Services routinely carry out around 670,000 fire safety check visits in England each year in people's homes. The aim of these 'Safe and Well Visits' is to reduce fire risks, support independent living, improve quality of life, and help prevent avoidable hospital admissions and excess winter deaths.

One part of the Safe and Well Visit is looking at ways to prevent falls. For some people, falling can cause serious health issues and in some cases may be fatal. About a third of people over the age of 65, and half of those over 80, will fall each year. Many of these falls happen at home. Falling may cause people to lose confidence, feel as if they have lost their independence and become withdrawn. About a fifth of all of the falls people have need medical attention. There were around 210,000 people admitted to hospital, as an emergency, in England in 2016 due to having had a fall. It costs the National Health Service (NHS) about £2.3 billion a year to treat patients who fall. The problem is likely to get worse as people are living longer. What investigators do not know is whether Safe and Well Visits undertaken by members of the Fire and Rescue Service reduce falls and can improve health-related quality of life and if they are good value for money.

To find out if Safe and Well Visits reduce the number of falls older people have and improve their quality of life, investigators will conduct a trial. The investigators will recruit 1156 people aged 70 years and over from lists of people held on Fire and Rescue Service databases or by advertising for participants and allocate half of the people to receive a Safe and Well Visit at the start of the study. The visit will last about an hour and will be tailored to the risks of the people living in the household. The other half of the people will receive the Safe and Well Visit after 12 months (when they have finished the study). Everyone will receive a falls prevention leaflet from Age United Kingdom and their usual care from their General Practitioner and other health care professionals. Participants will be asked to fill in monthly falls calendars and three postal questionnaires over 12 months to collect information about falls, their quality of life, how often they have used NHS services, and whether they are doing any activities that make them more likely to have a fire in their home. This information may be collected over the phone or investigators may send questionnaires in the post. Researchers will analyse the data to find out if the Safe and Well Visits reduce falls and if they are good value for money. The investigators also want to find out if the Safe and Well Visits are acceptable to older people and to the Fire and Rescue Service. This will be explored through a series of in-depth interviews. The investigators will assess treatment fidelity using the following strategies: observations of those delivering the Safe and Well Visits; delivery inventory will be completed for each participant; participant outcome questionnaires will include information on adherence with the intervention; and interviews with trial participants and members of the Fire and Rescue Service who delivered the Safe and Well Visits.

In addition to the main FIREFLI study investigators will undertake two additional trial methodological Studies within a Trial (SWAT) to evaluate one recruitment and one retention strategy. The first will test if using a recruitment invitation letter informed by Self-Determination Theory will increase the number of participants who take part in the study. The second will test if including a pen with the reminder four-month questionnaire will increase the number of postal questionnaires returned to the study team.

Once the trial is completed, the investigators will make sure the results can be used by as many people as possible. They will send the people who took part in the study a summary of the findings, and the results will be presented at relevant conferences and published in scientific journals. Investigators will share these findings with other Fire and Rescue Services.

ELIGIBILITY:
Main FIREFLI trial

Inclusion Criteria:

* Men and women aged 65 years and over in the Humberside FRS area or aged 79 and over in the Kent Fire and Rescue Service (FRS) area
* Community dwelling
* Willing to receive a SWV from the FRS

Exclusion Criteria:

* Living in a residential or nursing home
* Bed bound
* Unable to give informed consent to take part in the study and living alone
* Had an occupational therapist (OT) visit within the past 12 months
* Received a SWV from the FRS in the past three years
* Have been referred to the FRS as an urgent referral

For those participants who have been sent a recruitment pack directly from York Trials Unit (YTU) in response to advertising or hearing about the study, as opposed to receiving an invitation and recruitment pack via the mail out from the FRS, a further eligibility check is required to see if the participant is eligible for a Safe and Well Visit by the FRS. In these circumstances, there is another exclusion criterion: Not eligible for a Safe and Well Visit with the FRS.

Recruitment Study within a trial (SWAT)

Inclusion criteria Any patient identified by the Fire and Rescue Service as eligible to receive a FIREFLI trial invitation pack.

Retention SWAT Inclusion criteria For logistical reasons, all participants due to be sent a four month questionnaire will be randomised into the SWAT. However, only those sent a four month questionnaire reminder letter will be included in the analysis.

Exclusion criteria Participants who withdraw from follow-up before their four month questionnaire is due and those for whom it is not necessary to send a reminder letter will be excluded from the SWAT.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cockayne, Principal Investigator — University of York
Locations (2):
- United Kingdom (2):
  - Humberside Fire and Rescue Service, Hull, East Yorkshire
  - Kent Fire and Rescue Service, Maidstone, Kent

IPD SHARING:
Plan to Share IPD: No
Study data and resources to be shared with researchers upon request. Please contact at given details.

REFERENCES:
- [Derived] Cockayne S, Fairhurst C, Cunningham-Burley R, Mann J, Stanford-Beale R, Hampton S, Wilkinson S, Adamson J, Crossland S, Drummond A, Hewitt CE, Pighills A, Roberts G, Ronaldson S, Scantlebury A, Torgerson DJ; FIREFLI team. Effectiveness of Safe and Well Visits in reducing falls and improving quality of life among older people: The FIREFLI RCT. Public Health Res (Southampt). 2025 Sep;13(7):1-62. doi: 10.3310/DJHF6633. PMID 41013989
- [Derived] Adamson J, Scantlebury A, Drummond A, Fairhurst C, Cockayne S; Firefli team. Why do common sense trials fail in the UK? Lessons learned from a trial which tested the effectiveness and cost-effectiveness of a community falls prevention programme (the Firefli study). Trials. 2025 Sep 26;26(1):365. doi: 10.1186/s13063-025-09116-x. PMID 41013512
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- See also: National Institute of Health Research (NIHR) — https://www.fundingawards.nihr.ac.uk/award/NIHR128341
- See also: York Trials Unit, University of York, United Kingdom — https://www.york.ac.uk/healthsciences/research/trials/ytutrialsandstudies/archive/firefli/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants recruited to the recruitment Study within a Trial (SWAT) are the same participants as those in the main trial. They are not in addition to those recruited.
Groups:
- SWAT Intervention: Participants received an study invitation letter based on Self-Determination Theory
- SWAT Control Group: Participants received a study invitation letter based on 'standard' invitation letter sent out by the York Trials Unit
- Retention SWAT Intervention Arm: Participants due to be allocated to this arm were due to be sent a pen with their follow up questionnaire.
- Retention SWAT Control Group: Participants who were due to be allocated to this arm were not due to be sent a pen.
Period: Main FIREFLI Trial
Arm/Group | SWAT Intervention | SWAT Control Group | Main FIREFLI Trial: Intervention Arm | Main FIREFLI Trial: Control Arm | Retention SWAT Intervention Arm | Retention SWAT Control Group
Started | 0 | 0 | 32 | 31 | 0 | 0
Completed | 0 | 0 | 32 | 31 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Recruitment SWAT
Arm/Group | SWAT Intervention | SWAT Control Group | Main FIREFLI Trial: Intervention Arm | Main FIREFLI Trial: Control Arm | Retention SWAT Intervention Arm | Retention SWAT Control Group
Started (63 participants took part. These participants took part in the main trial but also in an embedded methodological substudy - recruitment Study within a Trial (SWAT). Participants were initially randomised to receive 1 of 2 invitation letters to take part in the study - 37 were allocated to the SWAT intervention and 26 to the SWAT control group. Participants were then randomised to the main FIREFLI trial - 32 to intervention and 31 to control. The periods therefore represent different studies.) | 37 | 26 | 0 | 0 | 0 | 0
Completed | 37 | 26 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SWAT Intervention: Participants received a study invitation letter based on Self-Determination Theory
- Total: Total of all reporting groups
Arm/Group | Main FIREFLI Trial: Intervention Arm | Main FIREFLI Trial: Control Arm | SWAT Control Group | SWAT Intervention | Total
Number analyzed (Participants) | 32 | 31 | 25 | 37 | 125
Age, Categorical [Count of Participants; unit: Participants] — Population: The main FIREFLI trial and the SWAT are two separate studies involving the same participants.
  Participants
    Main FIREFLI trial: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    Main FIREFLI trial: <=18 years | 0 | 0 | 0 | 0 | 0
    Main FIREFLI trial: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
    Main FIREFLI trial: >=65 years | 32 | 31 | 0 | 0 | 63
    SWAT trial: number analyzed (Participants) | 0 | 0 | 25 | 37 | 62
    SWAT trial: <=18 years | 0 | 0 | 0 | 0 | 0
    SWAT trial: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
    SWAT trial: >=65 years | 0 | 0 | 25 | 37 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: The main FIREFLI trial and the SWAT are two separate studies involving the same participants.
  years
    Main FIREFLI trial: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    Main FIREFLI trial | 80.6 (6.1) | 76.3 (4.0) |  |  | 78.5 (5.6)
    SWAT trial: number analyzed (Participants) | 0 | 0 | 25 | 37 | 62
    SWAT trial |  |  | 78.5 (6.0) | 78.5 (5.5) | 78.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: The main FIREFLI trial and the SWAT are two separate studies involving the same participants.
  Participants
    Main FIREFLI trial: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    Main FIREFLI trial: Female | 20 | 11 |  |  | 31
    Main FIREFLI trial: Male | 12 | 20 |  |  | 32
    SWAT trial: number analyzed (Participants) | 0 | 0 | 25 | 37 | 62
    SWAT trial: Female |  |  | 9 | 21 | 30
    SWAT trial: Male |  |  | 16 | 16 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Measure Analysis Population Description: The main FIREFLI trial and the SWAT are two separate studies involving the same participants - all from the UK.
  participants
    United Kingdom: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    United Kingdom | 32 | 31 |  |  | 63
EQ5D-5L (5 level EQ-5D) utility index value [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D-5L comprises 5 dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), each with 5 responses (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=unable to do/extreme problems), which lead to 3125 unique combinations of health states (e.g. 34221). Each health state is mapped to a utility index score on a scale from -0.59 to 1, where negative values correspond to a state worse than death, 0 corresponds to a health state equivalent to being dead and 1 corresponds to perfect health. Population: Measure Analysis Population Description: The main FIREFLI trial and the SWAT are two separate studies involving the same participants.
  units on a scale
    Main FIREFLI trial: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    Main FIREFLI trial | 0.724 (0.203) | 0.718 (0.252) |  |  | 0.721 (0.227)
    SWAT trial: number analyzed (Participants) | 0 | 0 | 25 | 37 | 62
    SWAT trial |  |  | 0.748 (0.243) | 0.707 (0.218) | 0.724 (0.227)
Fallen in past 12 months [Mean (Standard Deviation); unit: Number of falls] — Population: Measure Analysis Population Description: The main FIREFLI trial and the SWAT are two separate studies involving the same participants.
  Number of falls
    Main FIREFLI trial: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    Main FIREFLI trial | 0.88 (1.50) | 0.77 (1.92) |  |  | 0.83 (1.71)
    SWAT trial: number analyzed (Participants) | 0 | 0 | 25 | 37 | 62
    SWAT trial |  |  | 1.36 (2.25) | 0.49 (0.84) | 0.84 (1.72)
EQ5D-5L (5 level EQ-5D) VAS [Mean (Standard Deviation); unit: units on a scale] — The visual analogue scale (VAS) records participants' overall evaluation of their health on a scale from 0 (worst imaginable health) to 100 (best imaginable health) Population: Measure Analysis Population Description: The main FIREFLI trial and the SWAT are two separate studies involving the same participants.
  units on a scale
    Main FIREFLI trial: number analyzed (Participants) | 32 | 31 | 0 | 0 | 63
    Main FIREFLI trial | 75.8 (19.1) | 73.3 (20.7) |  |  | 74.6 (19.8)
    SWAT trial: number analyzed (Participants) | 0 | 0 | 25 | 37 | 62
    SWAT trial |  |  | 75.8 (19.2) | 74.1 (20.5) | 74.8 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Main FIREFLI Trial: The Number of Self-reported Falls Per Participant Over the 12 Months From Randomisation.
Description: The number of self-reported falls per participant over the 12 months from randomisation. A fall is defined as an unexpected event in which the participant comes to rest on the ground, floor, or lower level". Data will be collected prospectively via participant-reported monthly falls calendars.
Time Frame: Falls per participant over the 12 months from randomisation.
Population: Analysis not undertaken as followup data not collected
Arm/Group | Main FIREFLI Trial: Intervention Arm | Main FIREFLI Trial: Control Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Health-related Quality of Life Measured by the EuroQol 5 Dimensions, 5 Level Version
Description: Health-related self reported quality of life measured by the EuroQol 5 Dimensions. It measures health (functioning) in terms of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, respondents state whether they have no problems, slight problems, moderate problems, severe problems, or are unable to perform the activity. The EQ5D-5L will be used to calculate a EQ-5D-5L utility index score. A utility index score of one represents full health and a score of zero represents death, with it also being possible to have states worse than death as indicated by negative scores. A score of 1 is the best health and -0.574 the worst.
Time Frame: Over the 12 months from randomisation.
Population: Analysis not undertaken as followup data not collected.
Arm/Group | Main FIREFLI Trial: Intervention Arm | Main FIREFLI Trial: Control Arm
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Recruitment SWAT: Recruitment to the FIREFLI Trial.
Description: The proportion of participants randomised into the main FIREFLI trial calculated as the number of participants randomised to the main FIREFLI trial divided by the total number of recruitment packs mailed out to potential participants.
Time Frame: End of recruitment - approximately one year.
Measure: Count of Participants; unit: Participants
Arm/Group | SWAT Intervention | SWAT Control Group
Number analyzed (Participants) | 37 | 25
Participants | 37 | 25

4. Primary Outcome: Retention SWAT: Four-month Questionnaire Response Rate.
Description: The proportion of four-month reminder questionnaires returned to the York Trials Unit (YTU) calculated as the number of returned four-month follow-up questionnaires divided by the total number of four-month questionnaires mailed out to participants.
Time Frame: Four months from randomisation.
Reporting Status: Not Posted

5. Primary Outcome: The EuroQol-5D Visual Analogue Scale
Description: The EuroQol-5D Visual Analog Scale (VAS) score is a patient self-reported validated instrument. It consists of a vertical VAS with values between 0 (worst imaginable health) and 100 (best imaginable health), on which participants provide a global assessment of their health. Higher score indicate better health state.
Time Frame: Over 12 months since randomisation
Reporting Status: Not Posted

6. Secondary Outcome: Time to First Fall and Between Subsequent Falls.
Description: Time to each fall, with censoring at date of withdrawal, death or end of 12 month follow-up measured using fall data from monthly falls calendars or follow-up questionnaires. The time to the first fall will be derived as the number of days from randomisation until the patient reports having a fall. Time in days between any subsequent falls will also be calculated.
Time Frame: Over the 12 months from randomisation.
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Participants Reporting at Least One Fall.
Description: Proportion of participants reporting at least one fall in the 12 months from randomisation calculated as the number who report at least one fall on their monthly falls calendars or participant follow-up questionnaires divided by the total number of randomised participants.
Time Frame: Over the 12 months from randomisation.
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Participants Reporting Two or More Falls.
Description: Proportion of participants reporting at least two falls in the 12 months from randomisation calculated as the number who report at least one fall on their monthly falls calendars or participant follow-up questionnaires divided by the total number of randomised participants.
Time Frame: Over the 12 months from randomisation.
Reporting Status: Not Posted

9. Secondary Outcome: Fear of Falling
Description: Participants will be asked to score how often they have worried about falling in the past four weeks. Six response categories will be used (all of the time, most of the time, a good bit of the time, some of the time, a little of the time, and none of the time). This will be scored from a minimum of 1 to a maximum of 6 respectively and treated as continuous data. Minimum score is 1 and maximum score is 6, with higher scores indicating less concern about falling.
Time Frame: At four, eight and 12 months post-randomisation measured by asking participants to score how often they have worried about having a fall in the past four weeks.
Reporting Status: Not Posted

10. Secondary Outcome: Universtiy of California Los Angeles (UCLA) 3-item Loneliness Scale
Description: The UCLA 3-item loneliness scale is a screening tool for loneliness in adults. The scale consists of three questions that measure three dimensions of loneliness: relational connectedness, social connectedness, and self-perceived isolation. Each question is rated on a 3-point scale ('hardly ever' = 1 point, 'some of the time' = 2 points, 'often' = 3 points). The scores for each individual question are added together to give a possible range of scores from 3 to 9. A higher scores indicates a higher degrees of loneliness.
Time Frame: At four, eight and 12 months post-randomisation.
Reporting Status: Not Posted

11. Secondary Outcome: Fall Related Injuries and Costs.
Description: Fall-related injuries and costs over the 12 months from randomisation measured using participant self-reported data from follow-up questionnaires at four, eight and 12 months post-randomisation. The following data will be collected: injuries, healthcare resource use in primary care and community (i.e. General Practitioner, occupational therapist and physiotherapist) and secondary care (i.e. inpatient nights in hospital, day case attendances, outpatient attendances, and accident and emergency). Data on participant's time and expenses (i.e. travel costs and additional equipment) and informal care provided by friends/family, including productivity losses, will also be collected.
Time Frame: At four, eight and 12 months post-randomisation.
Reporting Status: Not Posted

12. Secondary Outcome: Fire Risk Taking Behaviours
Description: Fire risk taking behaviours measured using participant self-report.
Time Frame: At four, eight and 12 months post-randomisation.
Reporting Status: Not Posted

13. Secondary Outcome: Uptake of Flu Jab
Description: Uptake of flu jab using participant self-reported flu vaccination within the past 12 months.
Time Frame: Over the 12 months from randomisation.
Reporting Status: Not Posted

14. Secondary Outcome: Smoking/Vaping Status of Residents Within the Property
Description: Smoking/vaping status of residents within the property, smoking or vaping inside the property, smoking in bed, and referral to National Health Service stop smoking services at four, eight and 12 months measured using participant self-reported data from follow-up questionnaires at four, eight and 12 months.
Time Frame: At four, eight and 12 months post-randomisation.
Reporting Status: Not Posted

15. Secondary Outcome: Participant Reported Fire Within the Property That the FRS Attended at Four, Eight and 12 Months Post-randomisation.
Description: Participant reported fire within the property that the FRS attended at four, eight and 12 months post-randomisation
Time Frame: At four, eight and 12 months post-randomisation.
Reporting Status: Not Posted

16. Secondary Outcome: Participant Reported Fire Within the Property That Did Not Require the FRS to Attend.
Description: Fire incident.
Time Frame: At four, eight and 12 months post-randomisation.
Reporting Status: Not Posted

17. Secondary Outcome: Attendances to Participants' Homes for Fire Related Incidents as Recorded by the FRS.
Description: Fire incident.
Time Frame: At four, eight and 12 months post-randomisation..
Reporting Status: Not Posted

18. Secondary Outcome: Recruitment SWAT: Proportion of Participants Who Return a Screening Form
Description: Proportion of participants who return a screening form calculated as the number of participant-completed screening forms returned to YTU divided by the number of screening forms posted out to potential participants.
Time Frame: Enrollment
Reporting Status: Not Posted

19. Secondary Outcome: Recruitment SWAT: Proportion of Participants Who Are Eligible for Randomisation
Description: Proportion of participants who are eligible for randomisation calculated as the number of participants assessed as eligible for randomisation by researchers at YTU divided by the number of screening forms posted out to potential participants.
Time Frame: Enrollment
Reporting Status: Not Posted

20. Secondary Outcome: Recruitment SWAT: Retention in the Trial at Three Months Post-randomisation
Description: Proportion of participants who remain in the trial at three months post-randomisation calculated as the number of participants who return at least the first three months' worth of falls calendars from the date of randomisation, divided by the number of screening forms posted out to potential participants. This will also be calculated as a proportion of randomised participants.
Time Frame: Three months post-randomisation.
Reporting Status: Not Posted

21. Secondary Outcome: Retention SWAT: Time to Response
Description: Time to response calculated as the number of days between the four-month questionnaire being mailed out to the participant and the questionnaire recorded as being returned to York Trials Unit measured using the date the four-month questionnaire was mailed out and received back at YTU.
Time Frame: Four months post-randomisation.
Reporting Status: Not Posted

22. Secondary Outcome: Retention SWAT: Completeness of Response
Description: The number of completed questions on the four month questionnaire.
Time Frame: Four months post-randomisation.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study. The start of the adverse event reporting period for each participant was from the date the participant gave consent to be in the study. Adverse events were due to be collected over the 12 month duration the participant was in the study.
Description: Only serious adverse events reportable to the regulatory body Health Research Authority (https://www.hra.nhs.uk/), were reportable on this study.
Arm/Group | Main FIREFLI Trial: Intervention Arm | Main FIREFLI Trial: Control Arm | SWAT Intervention | SWAT Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/37 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/37 | 0/26
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/37 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT04717258/Prot_SAP_000.pdf